CLINICAL TRIAL: NCT05379452
Title: Outcomes of Neonates Born to Mothers With SARS-CoV-2 Infection During the Outbreak of Omicron in Shanghai: a Cohort Study.
Brief Title: Outcomes of Neonates Born to Mothers With SARS-CoV-2 Infection in Shanghai
Status: Terminated | Type: Observational
Why Stopped: The study was concluded as planned upon reaching its predetermined endpoint, which included the completion of data collection and achievement of the necessary sample size for statistical significance.
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_COVID19-2
Record Dates: First submitted 2022-05-16; First posted 2022-05-18 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: SARS-CoV2 Infection; Neonatal Infection; Outcomes
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Since March 2022, there are an outbreak of SARS-CoV-2 infection (Omicron) in Shanghai. This cohort study aims to analysis the clinical outcomes of neonates born to mothers with SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born to mothers with SARS-CoV-2 infections.

Exclusion Criteria:

* Parents who rejected to participate in this study.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates born to mothers with SARS-CoV-2 infections will be recruited from all the designated hospital during the outbreak of Omicron in Shanghai.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
The death of newborns | The date of discharge，an average of 4 weeks after the admission

SECONDARY OUTCOMES:
The malformation rate of neonates born to mothers with SARS-CoV-2 infections | Birth
The preterm delivery rate of neonates born to mothers with SARS-CoV-2 infections | Birth
The brain injury rate of neonates born to mothers with SARS-CoV-2 infections | within 7days after the admission
The development delay rate of neonates born to mothers with SARS-CoV-2 infections | within 1 year after the admission
The Chinese standardized Denver Developmental Screening Test (DDST) in neonates born to mothers with SARS-CoV-2 infections | Infants ( ≥35 weeks）are at 1 year after birth;Infants（< 35weeks） are at a corrected age of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes